CLINICAL TRIAL: NCT04163497
Title: Patient Experience: ICU Diaries and Its Effects After the Unit Discharge
Brief Title: ICU Diaries and Its Effects After the Unit Discharge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Ernesto Dornelles (Other)
Responsible Party: Principal Investigator, Juliana Mara Stormovski de Andrade, Principal Investigator, Hospital Ernesto Dornelles
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 3.011.427
Record Dates: First submitted 2019-07-31; First posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Post Intensive Care Unit Syndrome; Intensive Care Unit Syndrome; PTSD; Anxiety Symptoms; Depressive Symptoms
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The finaly analysis, by the statistician will be masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diary reading (Experimental)
  Interventions: Device: ICU Diaries
- No diary reading (No Intervention)

INTERVENTIONS:
Device: ICU Diaries — To explore the effects of providing an ICU Diary in the symptoms of anxiety, depression and PTSD within patients who were hospitalized in the unit.
  Arms: Diary reading

SUMMARY:
The preparation of ICU Diary, conducted by the Hospital care team towards the patient, has been suggested as an effective and low-cost strategy to enhance the patient's experience in the intensive care unit, as well as to prevent anxiety, depression and Posttraumatic Stress Disorder (PTSD). New-found researches in Brazilian ICUs indicates the pervasiveness of these symptoms in patients who have been hospitalized in the unit, however, there are no randomized trials that evaluate the impact of Diaries in the Brazilian context. The aim is to explore the effects of providing an ICU Diary in the symptoms of anxiety, depression and PTSD within patients who were hospitalized in the unit. Refers to a randomized controlled trial that is being conducted in two ICUs in a general-purpose hospital in Porto Alegre, Brazil.

DETAILED DESCRIPTION:
The Diaries will be filled voluntarily by the professionals who provide the patient care - psychologists, nutritionists, nursing technicians, nurses, physicians and physiotherapists. In addition, the patient's family members who wish to participate and collaborate with the Diaries may ask anyone on the team to assist them. The Diaries will be available at the bedside and may be filled with objective and subjective data on the patient's clinical condition and daily evolution, as well as remarkable events. Examples of entries possibilities are messages, pictures, drawings, photographs, thoughts, sayings, and wishes. Photographic records aim to provide the patient memories of the environment and of his advances in treatment. They will be attached to the Diary only if the patient wishes.

The predicted sample is composed of 102 intensive care patients, aged above 18 years old, that require mechanical ventilation and remained in the ICU more than 72 hours.

All patients who meet the inclusion criteria will have their Diary drawn up by the team and will be randomized one week after discharge from the ICU. All patients will have their memory assessed at 1 week deadline after critical care discharge, and at this moment, the intervention patients will receive their ICU Diary along with psychological support. One month after the ICU discharge, all the patients will be evaluated by phone and checked in symptoms of depression, anxiety and Posttraumatic Stress Disorder (PSTD).

The final assessment of the development of the symptoms will be at the deadline of 3 months.The patients in the control group will be invited to withdraw their Diary after the end of the survey. In case of readmission in the ICU, in a period less than 72h of discharge, the Diary used will be reactivated. In cases of death, the researchers will offer the responsible parent the opportunity to receive the Diary. During this period, the Diaries will be stored by the researchers confidentially, in a previously defined location.

ELIGIBILITY:
Inclusion Criteria:

* Will be included in this study ICU patients, older than 18 years old who are on mechanical ventilation, whose family members accept the participation by signing the consent form.

Exclusion Criteria:

* remain in the ICU for less than 72 hours;
* require mechanical ventilation for less than 24 hours;
* have limiting neurological symptoms (such as previous dementia);
* have a diagnosis of PTSD prior to hospitalization;
* have severe cognitive impairment at ICU discharge;
* not participate in all stages of the study, or whose outcome is death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-03-09 (Estimated); Study Completion 2020-09-09 (Estimated)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder (PTSD) | 1 week after ICU discharge
  number of patients with PTSD assessed by Posttraumatic Stress Disorder Checklist (PCL-5) - PCL-5
  A 20-item selfreport measure designed to assess the DSM-5 symptoms of PTSD. Responders are asked to rate how bothered they have been by each item in the past month on a 5-point Likert scale ranging from 0-4. A provisional PTSD diagnosis can be made by treating each item rated as 2 = "Moderately" or higher as a symptom endorsed, then following the DSM-5 diagnostic rule which requires at least: 1 Criterion B item (questions 1-5), 1 Criterion C item (questions 6-7), 2 Criterion D items (questions 8-14), 2 Criterion E items (questions 15-20). According the authors, a PCL-5 cut-point of 33 it's a reasonable value to use for provisional PTSD diagnosis.
Posttraumatic Stress Disorder (PTSD) | 1 month after ICU discharge
  number of patients with PTSD assessed by Posttraumatic Stress Disorder Checklist (PCL-5) - PCL-5
  A 20-item selfreport measure designed to assess the DSM-5 symptoms of PTSD. Responders are asked to rate how bothered they have been by each item in the past month on a 5-point Likert scale ranging from 0-4. A provisional PTSD diagnosis can be made by treating each item rated as 2 = "Moderately" or higher as a symptom endorsed, then following the DSM-5 diagnostic rule which requires at least: 1 Criterion B item (questions 1-5), 1 Criterion C item (questions 6-7), 2 Criterion D items (questions 8-14), 2 Criterion E items (questions 15-20). According the authors, a PCL-5 cut-point of 33 it's a reasonable value to use for provisional PTSD diagnosis.
Posttraumatic Stress Disorder (PTSD) | 3 months after ICU discharge
  number of patients with PTSD assessed by Posttraumatic Stress Disorder Checklist (PCL-5) - PCL-5
  A 20-item selfreport measure designed to assess the DSM-5 symptoms of PTSD. Responders are asked to rate how bothered they have been by each item in the past month on a 5-point Likert scale ranging from 0-4. A provisional PTSD diagnosis can be made by treating each item rated as 2 = "Moderately" or higher as a symptom endorsed, then following the DSM-5 diagnostic rule which requires at least: 1 Criterion B item (questions 1-5), 1 Criterion C item (questions 6-7), 2 Criterion D items (questions 8-14), 2 Criterion E items (questions 15-20). According the authors, a PCL-5 cut-point of 33 it's a reasonable value to use for provisional PTSD diagnosis.

SECONDARY OUTCOMES:
Anxiety | 1 week, 1 month and 3 months after ICU discharge
  number of patients with anxiety symptoms assessed by Hospital Anxiety and Depression Scale (HADS) - A self-assesment scale composed of 14 items rated on a 4-point Likert scale ranging from 0 to 3, with 5 of the 14 items reversed scored. Items from each of the 7-item anxiety and depression subscales are summed to give total subscale scores ranging from 0 to 21, with higher scores indicating higher levels of anxiety and depression.The cutoff points suggested by the authors were adopted: no anxiety from 0 to 8, with anxiety ≥ 9; no depression from 0 to 8, with depression ≥ 9.
Depression | 1 week, 1 month and 3 months after ICU discharge
  number of patients with depression symptoms assessed by Hospital Anxiety and Depression Scale (HADS) - A self-assesment scale composed of 14 items rated on a 4-point Likert scale ranging from 0 to 3, with 5 of the 14 items reversed scored. Items from each of the 7-item anxiety and depression subscales are summed to give total subscale scores ranging from 0 to 21, with higher scores indicating higher levels of anxiety and depression.The cutoff points suggested by the authors were adopted: no anxiety from 0 to 8, with anxiety ≥ 9; no depression from 0 to 8, with depression ≥ 9.

CONTACTS AND LOCATIONS:
Locations (1):
- Juliana Mara Stormovski de Andrade, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided